CLINICAL TRIAL: NCT01764295
Title: Multi-institutional, Randomized, Double-Blind, Placebo-Control, Factorial Design, 4-arms, 8 Week Administration, Phase 3 Clinical Study for Patients With Hypertension Associated With Dyslipidemia
Brief Title: Clinical Study for Patients With Hypertension Associated With Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: DW_DWJ1276003
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-01

CONDITIONS: Hypertension; Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — olmesartan; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- DWJ1276 (Experimental): Once daily, administered orally, 8 week
  Interventions: Drug: DWJ1276
- Olmesartan (Active Comparator): Once daily, administered orally, 8 week
  Interventions: Drug: Olmesartan
- Rosuvastatin (Active Comparator): Once daily, administered orally, 8 week
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator): Once daily, administered orally, 8 week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DWJ1276
  Arms: DWJ1276
Drug: Olmesartan
  Arms: Olmesartan
Drug: Rosuvastatin
  Arms: Rosuvastatin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of DWJ1276

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female in between ages of 20 and 80 at the time of screening
* Subject who can understand information provided and who can sign written consent voluntarily

Exclusion Criteria:

* Patients with hypersensitivity to olmesartan and rosuvastatin
* Pregnant or lactating women and fertile women who is not using proper contraceptive method
* Patient with history of drug or alcohol abuse

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
LDL-C percent change of DWJ1276 from baseline | 8weeks
DBP change of DWJ1276 from baseline | 8weeks

SECONDARY OUTCOMES:
Proportion of subjects who reached LDL-C treatment goal defined by NCEP ATP III guideline | 8weeks
Proportion of subjects who reached blood pressure treatment goal defined by JNC VII report | 8weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea